CLINICAL TRIAL: NCT01702103
Title: MULTICENTER, RANDOMIZED, DOUBLE BLIND, CONTROLLED, CLINICAL STUDY TO DEMONSTRATE THE THERAPEUTIC CLINICAL EQUIVALENCE OF TWO MOMETASONE NASAL SPRAYS IN THE RELIEF OF THE SIGNS AND SYMPTOMS OF PERENNIAL ALLERGIC RHINITIS.
Brief Title: Demonstrate the Therapeutic Clinical Equivalence of Two Mometasone Nasal Sprays
Acronym: PHT-01-12
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PH&T S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: PHT-01-12
Record Dates: First submitted 2012-09-12; First posted 2012-10-05 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Nasal Obstruction; Sneezing; Itching
MeSH Terms: conditions — Nasal Obstruction; Sneezing; Pruritus | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mometasone (Experimental): Mometasone, nasal spray for 8 weeks, 2 actuations each nostril in the morning.
  Interventions: Drug: Mometasone furoate
- Nasonex® (Active Comparator): Nasonex nasal spray for 8 weeks 2 actuations each nostril in the morning.
  Interventions: Drug: Mometasone furoate

INTERVENTIONS:
Drug: Mometasone furoate

SUMMARY:
Demonstrate the therapeutic clinical equivalence of two mometasone nasal sprays in the relief of the signs and symptoms of perennial allergic rhinitis, in term of changes at week 8 from baseline of Total Nasal Symptom Scores (TNSS).

DETAILED DESCRIPTION:
Perennial allergic rhinitis may be defined clinically as an inflammatory condition of the nose characterised by nasal obstruction, sneezing, itching, or rhinorrhoea. It occurs due to an exaggerated response to an environmental trigger which results in inflammation of the lining of the nose; it is similar to hayfever, however, the substances which cause the allergic reaction are present all year round; common causes include the faecal matter of the house dust-mite (Dermatophagoides pteronyssinus), animal proteins from domestic pets (saliva or skin proteins), and industrial dusts and fumes In those with perennial rhinitis, cigarette smoke, washing powders, detergents, strong perfume, and traffic fumes may exacerbate the condition.

According with WAO (World Allergy Organization), perennial rhinitis predominates in South America, Asia, Africa and Australia; perennial and seasonal rhinitis occur commonly in the U.S.A. and Japan. Seasonal rhinitis predominates in Europe. In one study in London of adults between the ages of 16 and 65 years, in 1991 the prevalence of rhinitis was 16%; of these, 8% had perennial symptoms, 6% perennial and seasonal symptoms, and 2% seasonal symptoms alone. As with asthma, both seasonal and perennial rhinitis seem to be increasing. The 2004-05 National Health Survey stated that 3.2 million Australians (approximately 16.1% of the population) self-reported experiencing symptoms of hay-fever and perennial rhinitis. The prevalence was found to be highest amongst those aged 25-34 and was slightly higher among females (1.7 million) than males (1.5 million).

Perennial allergic rhinitis (PAR) as seasonal allergic rhinitis (SAR) result from an immunological response mediated by IgE; there is also a Th2 cell component accounting for chronic symptoms. Histamine is a well-known mediator responsible for the signs and symptoms of SAR but many other mediators including leukotrienes and prostaglandin D2 are involved.

The management of perennial rhinitis involves the avoidance of triggers such as house dust-mite faeces and animal proteins, in conjunction with pharmacological treatments as:

Corticosteroids as Budesonide, Mometasone furoate, in the form of a nasal spray are the first-line treatment for perennial allergic rhinitis.

Antihistamines as Cetirizine hydrochloride, Fexofenadine hydrochloride, work by blocking the effects of histamine which is one of the main substances driving allergic reactions.

Decongestants as Phenylephrine hydrochloride, may be taken orally or as a nasal spray to reduce the secretions and swelling of the lining of the nose by constricting the blood vessels in the nose. Anti-inflammatories as Sodium cromoglycate, block the inflammatory pathways that cause the symptoms of perennial rhinitis, however, they have not been found to be more effective than corticosteroids or antihistamines.

Eye drops as Ketotifen fumarate, Hydrocortisone acetate, may be used to control symptoms such as itchy or watery eyes.

Allergen desensitisation involves exposing the patient to small doses of allergens in an attempt to desensitize them and prevent an allergic response.

Corticosteroids, as reported above, in the form of a nasal spray are the first-line treatment for perennial allergic rhinitis; one of the most widely used is mometasone furoate. A meta-analysis of randomized, double blind, placebo controlled, clinical trials on mometasone furoate nasal spray in the treatment of allergic rhinitis, by a comprehensive search of the MEDLINE, LILACS, SCOPUS, and the Cochrane Library databases up to 31 October, 2007 was carried out. Meta-analysis was performed with the random or the fixed effect models depending on heterogeneity, by using revman 5 software on the sixteen of the 113 identified articles that met the inclusion criteria. This meta-analysis provides a level Ia evidence for the efficacy of MFSN in the treatment vs placebo, with adverse events frequency similar in both groups.

On this basis we decided to design a trial to show therapeutic equivalence of a generic mometasone product with the drug Nasonex® Nasal Spray which is already marketed.

Number of patients: 298 completed patients with Perennial Allergic Rhinitis are required in this study; with a planned drop-out rate of 20%, 360 patients have to be enrolled.

Main Inclusion Criteria: Male and female, 12 years until 65 years old. Subjects with a minimum of 2 years of previous history of perennial allergic rhinitis to at least one perennial allergen at the time the study is being conducted.

Signed informed consent form. For patients under the age of majority the parent or legal guardian should sign the consent form and the child will be required to sign a patient "assent" form.

Subjects with perennial allergic rhinitis documented in writing positive allergic skin (a wheal >3mm) test or positive RAST test, performed at screening or within the past 12 months.

A score of at least 6 on the TNSS with a minimum score of at least 2 for "nasal congestion" and a minimum score of at least 2 for one of the remaining 3 symptoms.

Subjects capable of recording nasal allergy diary every day. Main Exclusion Criteria: Females who are pregnant, lactating or plan to get pregnant during the study.

History of asthma over the previous two years that required chronic therapy (with the exception of occasional acute or mild exercise induced asthma).

Patients with some nasal conditions (i.e. infectious sinusitis, hypertrophic rhinitis), or with clinically significant nasal deformity or any recent nasal surgery or trauma that has not completely healed.

Upper respiratory tract infection or any untreated systemic infections within the previous 30 days.

Patients previously treated with mometasone within the previous 30 days Patients who have received anti-allergy immunotherapy (desensitising subjects with increase of allergen challenges) in the previous 2 years or are still receiving this kind of therapy.

Patients with a history of tuberculosis. Patients with glaucoma, cataracts, ocular herpes simplex, conjunctivitis or other eye infection.

The patient has had recent exposure (30 days) or was at risk of being exposed to chicken pox or measles.

Any known hypersensitivity to mometasone, other steroids or any of the components of the study nasal spray.

Planned travel outside of the local area for more than 2 consecutive days or 3 days in total.

The patient has a history of alcohol or drug abuse.

ELIGIBILITY:
Inclusion Criteria:

Male and female, 12 years until 65 years old. Subjects with a minimum of 2 years of previous history of perennial allergic rhinitis to at least one perennial allergen at the time the study is being conducted.

Signed informed consent form. For patients under the age of majority the parent or legal guardian should sign the consent form and the child will be required to sign a patient "assent" form.

Subjects with perennial allergic rhinitis documented in writing positive allergic skin (a wheal >3mm) test or positive RAST test, performed at screening or within the past 12 months.

A score of at least 6 on the TNSS with a minimum score of at least 2 for "nasal congestion" and a minimum score of at least 2 for one of the remaining 3 symptoms.

Subjects capable of recording nasal allergy diary every day.

Exclusion Criteria:

Females who are pregnant, lactating or plan to get pregnant during the study. History of asthma over the previous two years that required chronic therapy (with the exception of occasional acute or mild exercise induced asthma).

Patients with some nasal conditions (i.e. infectious sinusitis, hypertrophic rhinitis), or with clinically significant nasal deformity or any recent nasal surgery or trauma that has not completely healed.

Upper respiratory tract infection or any untreated systemic infections within the previous 30 days.

Patients previously treated with mometasone within the previous 30 days Patients who have received anti-allergy immunotherapy (desensitising subjects with increase of allergen challenges) in the previous 2 years or are still receiving this kind of therapy.

Patients with a history of tuberculosis. Patients with glaucoma, cataracts, ocular herpes simplex, conjunctivitis or other eye infection.

The patient has had recent exposure (30 days) or was at risk of being exposed to chicken pox or measles.

Any known hypersensitivity to mometasone, other steroids or any of the components of the study nasal spray.

Planned travel outside of the local area for more than 2 consecutive days or 3 days in total.

The patient has a history of alcohol or drug abuse.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-01 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
demonstrate the therapeutic clinical equivalence of two mometasone nasal sprays in the relief of the signs and symptoms of perennial allergic rhinitis, in term of changes at week 8 from baseline of Total Nasal Symptom Scores (TNSS). | 8 weeks

SECONDARY OUTCOMES:
Safety monitoring AE, routine laboratory haematology, biochemical tests, urinalysis, assessment of adrenal function to be sure of lack of systemic effect of nasal spray formulation Overall Patient's and Physician's global assessment. | 8 weeks
  Patients at week 8 with a 50% reduction in TNSS mean change from baseline. Symptom-free days. The mean change from baseline to week 8 for mean Total Non Nasal Symptom Scores (TNNSS).
  Use of rescue medication (Time Frame: 8 weeks). Individual patient-rated symptoms evaluation. Clinical Global Improvement (CGI) evaluation.
  Treatment compliance:
  That includes description of the patient's adherence to the optimal prolonged treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Mazzetti, MD, Study Director — Sintesi Research Srl
Locations (1):
- Swiss Medical Group, Buenos Aires, Buenos Aires F.D., Argentina

REFERENCES:
- [Background] Sastre J, Mosges R. Local and systemic safety of intranasal corticosteroids. J Investig Allergol Clin Immunol. 2012;22(1):1-12. PMID 22448448